CLINICAL TRIAL: NCT05182944
Title: A Randomized, Controlled, Phase II Study of Perioperative Camrelizumab Combined With Albumin Paclitaxel and Cisplatin in Patients With Resectable Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Perioperative Camrelizumab Combined With Chemotherapy in Patients With Resectable ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Song Zhao, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L2021-Y346-002
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Cancer
Keywords: ESCC, perioperative, immune checkpoint inhibitor
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- After 2 cycles of neoadjuvant therapy,non-pCR patients adjuvant treatment (Experimental): After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, non-pCR patients adjuvant treatment（2-4 cycles Camrelizumab+Albumin Paclitaxel +Cisplatin and Camrelizumab maintenance treatment）
  Interventions: Drug: A：non-pCR patients
- non-pCR patients adjuvant treatment (Active Comparator): After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, non-pCR patients adjuvant treatment（Camrelizumab maintenance treatment）
  Interventions: Drug: B：non-pCR patients
- pCR patients adjuvant treatment (Experimental): After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, pCR patients adjuvant treatment（Camrelizumab maintenance treatment）
  Interventions: Drug: A：pCR patients
- pCR patients adjuvant treatment(BSC) (Active Comparator): After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, pCR patients adjuvant treatment（Best Supportive Care）
  Interventions: Drug: B：pCR patients

INTERVENTIONS:
Drug: A：non-pCR patients — After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, non-pCR patients adjuvant treatment（2-4 cycles Camrelizumab+Albumin Paclitaxel+Cisplatin and Camrelizumab maintenance treatment）
  Camrelizumab, 200 mg，Intravenous injection，q3W continuous medication Albumin Paclitaxel, 125 mg/m2, Intravenous injection d1,8 q3W continuous medication Cisplatin: 75mg/m2, Intravenous injection,d1, q3W continuous medication
  Arms: After 2 cycles of neoadjuvant therapy,non-pCR patients adjuvant treatment
Drug: B：non-pCR patients — After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, non-pCR patients adjuvant treatment（Camrelizumab maintenance treatment）
  Camrelizumab, 200 mg，Intravenous injection，q3W continuous medication Albumin Paclitaxel, 125 mg/m2, Intravenous injection d1,8 q3W continuous medication Cisplatin: 75mg/m2, Intravenous injection,d1, q3W continuous medication
  Arms: non-pCR patients adjuvant treatment
Drug: A：pCR patients — After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, pCR patients adjuvant treatment（Camrelizumab maintenance treatment）
  Camrelizumab, 200 mg，Intravenous injection，q3W continuous medication Albumin Paclitaxel, 125 mg/m2, Intravenous injection d1,8 q3W continuous medication Cisplatin: 75mg/m2, Intravenous injection,d1, q3W continuous medication
  Arms: pCR patients adjuvant treatment
Drug: B：pCR patients — After 2 cycles of neoadjuvant therapy（Camrelizumab+Albumin Paclitaxel+Cisplatin）, pCR patients adjuvant treatment（Best Supportive Care）
  Camrelizumab, 200 mg，Intravenous injection，q3W continuous medication Albumin Paclitaxel, 125 mg/m2, Intravenous injection d1,8 q3W continuous medication Cisplatin: 75mg/m2, Intravenous injection,d1, q3W continuous medication
  Arms: pCR patients adjuvant treatment(BSC)

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of camrelizumab combined with albumin paclitaxel and cisplatin as perioperative treatment of advanced esophageal squamous cell.

DETAILED DESCRIPTION:
The incidence of esophageal cancer is ranked seventh in the world, and the mortality rate ranks sixth in the world. Surgical treatment of early esophageal cancer has a good prognosis, and advanced esophageal cancer often requires a combination of surgery, chemotherapy, radiotherapy and immunotherapy, but the prognosis is still poor. The investigators designed a randomized, controlled, phase II study of perioperative camrelizumab combined with albumin paclitaxel and cisplatin in patients with resectable esophageal squamous cell carcinoma. The purpose of this study is to observe and evaluate the efficacy and safety of camrelizumab combined with albumin paclitaxel and cisplatin as perioperative treatment of advanced esophageal squamous cell.

ELIGIBILITY:
Inclusion Criteria:-

1. Aged 18-80 years, males or females；
2. Histologically or cytologically confirmed as ESCC；
3. Esophageal squamous cell carcinoma without anti-tumor treatment, and the clinical stage is T1b-2N+M0 or T3-4aN+/-M0 (AJCC/UICC TNM staging system 8th edition);
4. It can provide tumor tissue for the detection of PD-L1 expression level;
5. Follow-up surgery plan: radical esophageal squamous cell carcinoma surgery with esophagogastric reconstruction combined with at least complete 2 field lymph node dissection;
6. ECOG: 0~1;
7. Expected survival time ≥ 12 weeks;
8. Body mass index (BMI) ≥ 18.5kg/m2 or pg-sga score A / B;
9. 1）White blood cell count (WBC) ≥3.0 × 109/L, absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet (PLT) count ≥100×109/L, hemoglobin (HGB) ≥90 g/L, No blood transfusion or other hematopoietic factor treatment for the previous 14 days； 2）Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤2.5×upper limit of normal (ULN); serum total bilirubin (TBIL) ≤1.5×ULN ; Albumin (ALB) ≥30g/L; 3）Serum creatinine (CRE)≤1.0×ULN, creatinine clearance (Ccr)≥60 mL/min (Cockcroft-Gault formula); 4）International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) ≤ 1.5 × ULN;
10. Important organ functions: a) Heart function: normal or grade I; b) Lung function: FEV1>1.2L, FEV1% >40%; c) Liver function: Child-Pugh grade 5-6 points;
11. For premenopausal women (postmenopausal women must have been postmenopausal for at least 12 months to be considered infertile), the serum pregnancy test result is negative. Male subjects (including male subjects' female spouses of childbearing age) and female subjects of childbearing age must contraception from the first study drug administration to 6 months after the last study drug administration；
12. Obtain the informed consent signed by the subject or his legal representative;
13. Can cooperate to complete research procedures and follow-up inspections。

Exclusion Criteria:

1. Cervical esophageal squamous cell carcinoma;
2. Combined with cervical, supraclavicular, abdominal, retroperitoneal and pelvic lymph node metastasis (except pericardial lymph node metastasis and left gastric lymph node metastasis);
3. Previously received anti-tumor therapy for the primary disease (including surgery, chemotherapy, targeted therapy, immunotherapy, anti-angiogenesis therapy, radiotherapy, radiofrequency ablation, etc.) and other research treatments, except for Chinese patent medicines or Chinese herbal medicines stopped for more than 7 days ；
4. Previously received anti-tumor therapy for the primary disease (including surgery, chemotherapy, targeted therapy, immunotherapy, anti-angiogenesis therapy, radiotherapy, radiofrequency ablation, etc.) and other research treatments, except for Chinese patent medicines or Chinese herbal medicines stopped for more than 7 days ；
5. Previously active, potentially relapsed or undiagnosed autoimmune diseases, skin diseases (vitiligo, psoriasis, alopecia) without systemic treatment, well controlled type I diabetes, hypothyroidism (only thyroid hormone replacement therapy), and other diseases that were not expected to relapse under external stimulation were included.
6. History of allogeneic stem cell transplantation or organ transplantation;
7. Complicated with interstitial pneumonia or interstitial lung disease, non infectious pneumonia;
8. History of gastrointestinal perforation and/or fistula, abdominal abscess, visceral fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive within 6 months before the first study drug administration bowel resection (including partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea;
9. Major operations (except puncture and biopsy) or major trauma were performed ≤ 28 days before the administration of the first study drug;
10. Have vaccinated or plan to vaccinate live vaccine within 28 days before the first study drug administration;
11. Use corticosteroids (>10 mg/day prednisone or equivalent dose) or other immunosuppressive agents within 14 days before the first study drug administration. Inhalation, ophthalmic, intra-articular, intranasal or topical corticosteroids can be used prophylactically for short-term (≤7 days) use of corticosteroids (for example, to prevent allergy to contrast agents) or for the treatment of non-autoimmune conditions (for example, delayed hypersensitivity caused by contact with allergens)
12. Infectious diseases that affect activities of daily living or require systemic treatment (such as the use of hormones, antibiotics, antifungal drugs, antiviral drugs, and oxygen inhalation) within 14 days before the first study drug administration, including but not limited to the need Hospitalized infections, bacteremia, severe pneumonia, etc.;
13. Combined with the following diseases that have not been well controlled, such as: a) New York Heart Association (NYHA) ≥ Grade 2 heart failure, b) Severe/Unstable Angina, c) Myocardial infarction ≤ 6 months before study administration, d) Severe arrhythmia requiring medication or intervention, e) Uncontrollable hypertension, f) Occurrence/combined arterial and/or venous thromboembolism ≤2 months before the first study administration, g) ≤6 before the first study administration A cerebrovascular accident occurred within a month, h) diabetes that has not been effectively controlled, i) thyroid disease that has not been effectively controlled, j) urine protein ≥ 2+ and 24-hour urine protein quantification ≥ 1.0g;
14. Tuberculosis (TB) who has received anti-tuberculosis treatment within 1 year before receiving/receiving/first study administration;
15. Human immunodeficiency virus infection (HIV1/2 antibody positive);
16. Acute or chronic active hepatitis B and / or hepatitis C: positive for hepatitis B virus surface antigen (HBsAg) / positive for hepatitis B virus core antibody (HBcAb) and positive for hepatitis B virus DNA (HBV DNA >2000 IU/ml or 103 copies /ml), if HBsAg/HB cAb positive, HBV DNA less than 2000 IU/ml or 103 copies of /ml can be entered, but entecavir or other anti HBV drugs should be taken simultaneously; hepatitis C virus (positive) antibody is positive and HBV copies;
17. Pregnant or lactating women;
18. Complicated with other malignant tumors ≤5 years before the first study drug administration, various cancers in situ, skin basal cell carcinoma or squamous cell carcinoma that have been cured in the past, local prostate cancer after radical resection, and catheters after radical resection except for carcinoma in situ;
19. Combined with other severe, acute, chronic or mental illness that may increase the risk of study medication or may interfere with the interpretation of the study results, the presence of alcoholism, drug abuse, or drug abuse, and other conditions that are not conducive to study drug administration, drug toxicity or adverse events (AE) Circumstances that lead to a decrease in the compliance of research behavior;
20. Other circumstances that the researcher considers inappropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response，pCR | At time of surgery
  defined as the absence of any viable tumor at the time of surgical resection, as assessed by central and local pathology laboratory
3 years disease free survival, DFS | up to 3 year
  Time after R0 resection to disease recurrence or death

SECONDARY OUTCOMES:
Major pathological response（MPR） | At time of surgery
  defined as ≤ 10% residual viable tumor at the time of surgical resection, as assessed by central pathology laboratory.
Objective Response Rate (ORR) | up to 2 year
  CR（ complete response）+PR（partial response）
Disease-Free Survival (DFS) | up to 5 year
  Time after R0 resection to disease recurrence or death
Overall Survival (OS) | up to 5 year
  defined as the time from randomization to death from any cause during the course of the study.
European Organisation for Research and Treatment of Cancer （EORTC） Multi-trait scaling analyses and face validity refined the module to four scales and six single items (QLQ-OES18). | up to 5 year
  EORTC QLQ-OES18

OTHER OUTCOMES:
The exploration of biomarkers | up to 2 year
  Exploring circulating tumor cells and circulating tumor DNA in neoadjuvant immunotherapy and adjuvant therapy for esophageal squamous cell carcinoma application value in immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Song Zhao, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China